CLINICAL TRIAL: NCT03064828
Title: Colorectal Adenoma Screening by Low-dose CT Colonoscopy With Computer-aided Detection
Brief Title: Colorectal Polyps Screening With Low-dose CT Colonoscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Collaborators: Air Force Military Medical University, China (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: KY20162082-1
Record Dates: First submitted 2017-01-24; First posted 2017-02-27 (Actual); Last update posted 2018-07-20 (Actual); Status verified 2017-11

CONDITIONS: Polyps; Colorectal Neoplasm
MeSH Terms: conditions — Polyps; Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CT colonoscopy(normal dose) (Active Comparator): Perform CT colonoscopy with full bowel preparation and inflated colon, CT Scans on subjects with normal-dose protocol by setting scanning parameters as 120-140 kilovolts peak (kVp), 100-200mA
  Interventions: Radiation: CT colonoscopy(normal dose)
- CT colonoscopy(low dose) (Experimental): Perform CT colonoscopy with full bowel preparation and inflated colon, CT Scans on subjects with normal-dose protocol by setting scanning parameters as 120-140 kVp, 20-100mA
  Interventions: Radiation: CT colonoscopy (low dose)

INTERVENTIONS:
Radiation: CT colonoscopy(normal dose) — Perform CT colonoscopy with full bowel preparation and inflated colon,CT Scans on subjects with normal-dose protocol by setting scanning parameters as 120-140 kVp, 100-200mA
  Arms: CT colonoscopy(normal dose)
Radiation: CT colonoscopy (low dose) — Perform CT colonoscopy with full bowel preparation and inflated colon,CT Scans on subjects with normal-dose protocol by setting scanning parameters as 120-140 kVp, 20-100mA
  Arms: CT colonoscopy(low dose)

SUMMARY:
This preliminary clinical trial aims to evaluate the performance of the low-dose CT colonoscopy (CTC) with computer aided detection (CAD) on polyps detection compared with optical colonoscopy (OC), and explore the possible clinical routine for integrated use of CT colonoscopy and optical colonoscopy OC in colorectal cancer screening.

DETAILED DESCRIPTION:
CT colonoscopy (CTC), also referred to as virtual colonoscopy (VC), utilizes computer virtual-reality techniques to navigate inside a three-dimensional patient-specific colon model reconstructed from abdominal CT images, looking for colonic lesions, full bowel preparation and colon inflation are needed to perform CTC examination. The clinical trial consists of two major parts:

1. Comparative study on the performance of CTC and OC: 50 subjects will be recruited in this part with written consents. With full bowel preparation, all the volunteers receive CT scans first with inflated colon, then OC followed by the same day, and necessary pathological analysis thereafter. The performance of CTC based on high-resolution CT data, including the number of polyps detected, size, position, etc, will be validated by that of OC with the paired comparison.
2. Integrate use of low-dose CTC with OC for colorectal cancer screening: After the validation of CTC performance, in this part, another 50 subjects will be recruited to explore the integrated use of CTC with OC as a possible and efficient workflow for colorectal cancer screening. In this part, a combination of normal dose and low-dose scan protocols will be employed (e.g., normal dose on supine, low-dose on prone), low-dose CTC based on the low-dose CT scanning protocol and an artifacts reduction technique will be introduced to reduce the radiation risk in screening.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with gastrointestinal symptoms potentially suggestive of colorectal cancer, such as diarrhea, constipation, abdominal pain or discomfort, rectal bleeding, iron-deficiency anemia, and unintended weight loss.
* Subjects with pathological confirmed colorectal cancer or polyps that need follow-up examination.
* Subjects with written consents

Exclusion Criteria:

* Subjects with acute colitis
* Acute diverticulitis
* Inguinal hernia including colon
* Colorectal surgery or endoscopic biopsy or resection of polyps within 6 months
* Known or suspected as colon perforated
* Complete intestinal obstruction
* Pregnant or lactating women

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-01; Primary Completion 2018-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of low-dose CTC for the polyp detection | within the first 30 days (plus or minus 3 days) after the completion of the first part of the trial
  return the number of polyps detected by low-dose CTC for each participant, sensitivity and specificity of low-dose CTC for the polyp detection can be derive from it with OC results as reference.

SECONDARY OUTCOMES:
CT radiation | within the first 3 days after each examination.
  Record the dose-length product of each CT scan for CTC participants and radiation dose of each scan can be derived from it.
Sensitivity and specificity of CTC for the detection of polyps with different shapes | within the first 30 days after the completion of the trial.
  Return the shape and location information of polyps detected by OC and CTC for each participant to reflect the CTC performance for the detection of polyps with different morphologies, especially for three major morphologic categories: sessile, pedunculated, and flat.
Sensitivity and specificity of CTC for the detection of poly malignancy | within the first 30 days after the completion of the trial.
  Return the histological types of polyps biopsied through OC after pathologic examination to reflect the CTC performance for the detection of polyp malignancy, especially the capability to differentiate adenomatous polyps from hyperplastic polyps.

CONTACTS AND LOCATIONS:
Overall Officials: Shuhui Liang, MD, Study Director — Air Force Military Medical University, China; Jiang Meng, MS, Principal Investigator — Air Force Military Medical University, China; Xiaofeng Zhang, MD, Principal Investigator — Air Force Military Medical University, China; Hong Yin, MD, Principal Investigator — Air Force Military Medical University, China; Hainan Sang, MS, Principal Investigator — Air Force Military Medical University, China
Locations (1):
- Xi jing Hospital, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Undecided